CLINICAL TRIAL: NCT01041248
Title: Efficacy of Tocilizumab in a Patient With Relapsing Polychondritis
Brief Title: Single Patient Study to Treat Relapsing Polychondritis With Tocilizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Johannes Roth, Pediatric Rheumatologist, Children's Hospital of Eastern Ontario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 25245
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Relapsing Polychondritis
Keywords: Relapsing Polychondritis; Single Patient Study; Tocilizumab
MeSH Terms: conditions — Polychondritis, Relapsing | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tocilizumab (Experimental): Single arm open label study. In this arm patient will receive 8mg/kg of Tocilizumab q 2 weeks iv.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 8mg/kg every 2 weeks i.v.
  Other Names: Actemra

SUMMARY:
Relapsing polychondritis (RP) is a rare, immune-mediated disease associated with inflammation in cartilaginous structures and other tissues throughout the body. Prognosis can be poor, especially in cases where there is acute involvement of the laryngotracheal cartilages leading to airway destruction, which are resistant to treatments such as corticosteroids, immunosuppressive or cytotoxic drugs. The pathogenesis remains unclear although it is thought that autoimmune reactions to antigens present in cartilages, such as type II collagen and matrilin may evoke symptoms. There are no known clinical or laboratory measures that predict the expression of specific disease manifestations or the overall disease course. Two recently published case reports have shown an association with elevated serum IL-6 levels and relapsing polychondritis. In these case reports, both patients with refractory relapsing polychondritis were treated with tocilizumab, a humanized monoclonal antibody to the Interleukin 6 receptor, and achieved sustained response to the drug. This single patient trial aims to evaluate the response to Tocilizumab in an eight year old boy with relapsing polychondritis who has been shown to have elevated serum IL-6 levels and who has responded poorly to conventional therapies. The study hypothesis is that Tocilizumab will be able to control the disease in this patient.

DETAILED DESCRIPTION:
In this N = 1 study a single known patient with relapsing polychondritis who has failed methotrexate, various anti TNF medications, anti IL1 medication and prolongued glucocorticosteroids will be recruited to receive Tocilizumab 8 mg /kg q 2 weeks iv.

The objective is to assess efficacy of tociliuzmab in combination with stable ongoing therapy. Our patient received tocilizumab 8 mg/kg over 1 hour by intravenous infusion every 2 weeks throughout the course of the study. To assess tocilizumab efficacy, the primary objective is the change in physician global assessment on a 100-mm horizontal visual analogue scale (VAS) of disease activity.

The secondary objectives were the change in parent global assessment of disease activity on a 100 mm VAS and the glucocorticoid dose in mg per day. Frequency of adverse events was also measured at baseline and after each biweekly tocilizumab infusion.

ELIGIBILITY:
Inclusion Criteria:

* Refractory relapsing polychondritis
* Failed glucocorticoid and methotrexate therapy

Exclusion Criteria:

* This is an N=1 clinical trial with a known patient, therefore, exclusion criteria are non-applicable.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Roth, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Kawai M, Hagihara K, Hirano T, Shima Y, Kuwahara Y, Arimitsu J, Narazaki M, Ogata A, Kawase I, Kishimoto T, Tanaka T. Sustained response to tocilizumab, anti-interleukin-6 receptor antibody, in two patients with refractory relapsing polychondritis. Rheumatology (Oxford). 2009 Mar;48(3):318-9. doi: 10.1093/rheumatology/ken468. Epub 2008 Dec 23. No abstract available. PMID 19106169

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 1 (January 2010)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 10 [10 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment of Disease Activity
Description: Physician global assessment of disease activity was assessed on a 100 mm Visual Analogue Scale where 0 would be no disease activity and 100 would be the maximum disease activity. Higher values therefore indicate higher disease activity and therefore a worse outcome. Change of this outcome measure over time was documented.
Time Frame: Baseline and then every 2 weeks prior to each infusion for total duration of 30 weeks
Population: a known patient for whom this trial was designed was recruited into this open label single arm study
Measure: Number; unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
mm
  Baseline | 21
  2 weeks | 14
  4 weeks | 12
  6 weeks | 43
  8 weeks | 14
  10 weeks | 12
  12 weeks | 8
  14 weeks | 6
  16 weeks | 5
  18 weeks | 8
  20 weeks | 0
  22 weeks | 2
  24 weeks | 0
  26 weeks | 37
  28 weeks | 19
  30 weeks | 0

2. Secondary Outcome: Prednisone Dose
Description: Prednisone dose administered to patient reduction through treatment course
Time Frame: 30 weeks
Population: single arm open label study for 1 patient with relapsing polychondritis
Measure: Number; unit: mg
Groups:
- Tocilizumab: treatment arm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
mg
  Baseline | 25
  2 weeks | 25
  4 weeks | 25
  6 weeks | 25
  8 weeks | 25
  10 weeks | 30
  12 weeks | 30
  14 weeks | 30
  16 weeks | 30
  18 weeks | 30
  20 weeks | 25
  22 weeks | 25
  24 weeks | 25
  26 weeks | 20
  28 weeks | 20
  30 weeks | 20

3. Secondary Outcome: Parent/Patient Global Assessment of Overall Well Being
Description: A 100 mm visual analogue scale was used for the assessment of the parent/patient globale well being, maximum value is 100 and minimum value is 0 with lower values being better well being and therefore improved outcome and higher values worse well being and therefore worse outcome. Changes in this score over time are being assessed with this measure.
Time Frame: 30 weeks
Population: Patient receiving Tocilizumab
Measure: Number; unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
mm
  Baseline | 53
  2 weeks | 0
  4 weeks | 0
  6 weeks | 33
  8 weeks | 12
  10 weeks | 2
  12 weeks | 0
  14 weeks | 1
  16 weeks | 1
  18 weeks | 2
  20 weeks | 0
  22 weeks | 1
  24 weeks | 0
  26 weeks | 30
  28 weeks | 15
  30 weeks | 0

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No